CLINICAL TRIAL: NCT01218503
Title: The Neural Correlates of Food Choice Decision-making in Obesity and Weight Loss (CHOICES)
Brief Title: The Neural Correlates of Food Choice Decision-making in Obesity and Weight Loss
Acronym: CHOICES
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Miriam Hospital (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); California Institute of Technology (Other)
Responsible Party: Principal Investigator, Kathryn E. Demos, Assistant Professor (Research), The Miriam Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: BRAIN-T32; K01DK090445 (NIH)
Record Dates: First submitted 2010-10-07; First posted 2010-10-11 (Estimated); Last update posted 2013-07-29 (Estimated); Status verified 2013-07

CONDITIONS: Obesity; Weight Loss; Weight Control
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CHOICES - obese (Experimental): behavioral weight loss treatment - overweight/obese females
  Interventions: Behavioral: CHOICES - obese

INTERVENTIONS:
Behavioral: CHOICES - obese — Standard group behavioral weight loss treatment

SUMMARY:
This study is designed to determine whether obese, normal weight, and successful weight loss maintainers differ in their food choice decision-making and/or executive function, and whether participation in a behavioral weight loss program leads to neural and/or behavioral changes. The investigators will examine behavioral performance on several tasks involving decision-making and self-control in conjunction with brain imaging data acquired during a food-choice decision-making task. Participants enrolled in the behavioral weight loss program will also be assessed following the treatment.

ELIGIBILITY:
Inclusion Criteria:

* women, ages 35-55, who are either currently obese (BMI = 30-40 kg/m2), always normal weight (lifetime BMI < 25, NW) or successful weight loss maintainers who have lost 10% of their body weight and maintained that loss for at least 1 year (lifetime maximum BMI = 30-40 kg/m2)

Exclusion Criteria:

* weight loss medications, binge eating, standard MRI contraindications (e.g., metal implants, claustrophobia, pregnancy), left-handedness, food allergies, neurological or psychiatric conditions, including but not limited to schizophrenia, bipolar disorder, epilepsy, stroke and traumatic brain injury with loss of consciousness, and, among obese participants, inability to participate at two time points and lack of interest in participating in a behavioral weight loss trial
* serious current physical disease (e.g., heart disease and cancer) for which physician supervision of diet and exercise prescription is needed, physical problems that limit the ability to exercise, participation in a weight loss program in the last 2 months and intention to become pregnant in the next 6 months

Ages: 35 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2010-03; Primary Completion 2016-10 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
fMRI | pre- and post-treatment in obese group, single time point for SWLM and NW

SECONDARY OUTCOMES:
Behavioral data | pre- and post-treatment of obese group, single time point for SWLM and NW

CONTACTS AND LOCATIONS:
Locations (1):
- Weight Control & Diabetes Research Center, Providence, Rhode Island, United States